CLINICAL TRIAL: NCT06659328
Title: Influence of Rhythm and Interpersonal Relationship on Gait Parameters in Children with Autism Spectrum Disorder: a Controlled Intervention Study
Brief Title: Influence of Rhythm and Interpersonal Relationship on Gait Parameters in Children with Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Estrada Barranco, Principal investigator, Universidad Europea de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASD intervention
Record Dates: First submitted 2024-10-04; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; stability; interpersonal relationship; gait patterns; proprioception
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This study employs a single-group, quasi-experimental design, where 30 children aged 4 to 6 years with Autism Spectrum Disorder (ASD) participate in a structured walking intervention. The intervention consists of observing the children's gait parameters under varying conditions: walking at normal (120 bpm), slow (100 bpm), and fast (140 bpm) rhythms, while accompanied by either a familiar adult or an unfamiliar adult. Each child will walk a distance of 10 meters, with their gait parameters-such as stride length, step time, cadence, velocity, and joint amplitudes-measured using video analysis software (Kinovea©). This sequential approach enables the assessment of the impact of both speed and social interaction on gait dynamics in a controlled environment. The study aims to elucidate how these factors influence locomotion in children with ASD, providing insights for future therapeutic interventions and rehabilitation strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Walking Intervention with Varying Speeds and Social Interaction in Children with Autism Spectrum Dis (Experimental): This arm of the study focuses on a single group of participants consisting of 30 children aged 4 to 6 years diagnosed with ASD. The objective is to evaluate how varying walking speeds and social interactions influence gait parameters.
  Participants will engage in a structured walking intervention under three conditions: normal speed (120 bpm), slow speed (100 bpm), and fast speed (140 bpm). Each child will walk with two different types of adult companions: a familiar adult (e.g., caregiver) and an unfamiliar adult. This design allows for a comprehensive assessment of gait characteristics in response to different social contexts and pacing.
  Each child will complete a 10-meter walking task, with gait parameters such as stride length, step time, cadence, velocity, and joint amplitudes being recorded using video analysis software (Kinovea©).The results will contribute to understanding how children with ASD adapt their locomotion to social cues and varying speeds
  Interventions: Procedure: Structured Walking Intervention for Children with Autism Spectrum Disorder

INTERVENTIONS:
Procedure: Structured Walking Intervention for Children with Autism Spectrum Disorder — Participants: Thirty children with ASD will participate in the walking sessions.
  Conditions: Each child will walk under three different speed conditions:
  Normal Speed: 120 beats per minute (bpm) Slow Speed: 100 bpm Fast Speed: 140 bpm
  Social Interaction: Each child will walk with two different types of adult companions:
  Familiar Adult: A caregiver or individual known to the child. Unfamiliar Adult: An adult not known to the child. Procedure: The walking distance will be 10 meters. The adult will wear a metronome in an earbud to ensure that they maintain the prescribed walking speed, which the child will be instructed to follow. Each child will experience all combinations of walking speeds and social interactions, allowing for a comprehensive assessment of how these factors influence gait parameters.
  Gait Parameters: The following parameters will be recorded during each walking session using video analysis software (Kinovea©):
  Stride length Step time Cadence Velocity Joint amplitudes

SUMMARY:
Autism Spectrum Disorder (ASD) affects social communication and motor coordination, with less synchrony with others and atypical gait patterns. Relationship with the adult or speed modify gait parameters in children diagnosed with ASD between 4 and 6 years old. Methodology: a cross-sectional observational design was carried out. The aim of this study was to analyze gait pattern variations in children with ASD in different speed conditions and modifying the social environment.

DETAILED DESCRIPTION:
Study Design:

This is a quasi-experimental, cross-sectional study designed to assess the influence of rhythm and interpersonal relationships on gait parameters in children diagnosed with Autism Spectrum Disorder (ASD). The study involved 30 children, aged 4 to 6, diagnosed with ASD (level I or II), who demonstrated independent walking ability without assistive devices. The children were recruited from Fundación AMÁS, an early intervention center.

Intervention:

The study aimed to analyze the gait of children under three different speed conditions-normal (120 beats per minute), slow (100 beats per minute), and fast (140 beats per minute)-while walking alongside either a familiar adult or a stranger. The intervention involved the following steps:

Preparation: Each child was informed about the walking activity and the adult who would accompany them. They were instructed to walk alongside the adult for a distance of 10 meters.

Walking Conditions:

Walking with a Familiar Adult: Children walked alongside an adult they knew, maintaining the specified rhythm.

Walking with a Stranger: Children walked alongside an unfamiliar adult at the same designated rhythm.

Speed Variation: The rhythm was controlled using a metronome, which only the accompanying adult could hear. The adult was instructed to adjust their walking pace according to the specified rhythm while guiding the child.

Recording and Analysis: The walking sessions were recorded using a camera positioned at a lateral view, ensuring consistent height and distance. The central 2 meters of the 10-meter path were analyzed using Kinovea© software to assess gait parameters.

Outcome Measures:

The study sought to evaluate several dependent variables, including:

Stride Length: The distance covered with each step. Step Time: The duration of each step. Cadence: The number of steps taken per minute. Velocity: The speed of walking measured in meters per second. Joint Amplitudes: The angles at which the hip, knee, and ankle joints moved during each phase of the gait cycle.

Study Population:

The study included children with ASD who attended regular therapy sessions at Fundación AMÁS. Inclusion criteria required children to be between 4 and 6 years old, with a clinical diagnosis of ASD (level I or II), and the ability to walk independently. Exclusion criteria included any associated syndromes or recent lower-limb interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 6 years.
* Clinical diagnosis of Autism Spectrum Disorder (ASD) (Level I or II).
* Ability to walk independently without the use of assistive devices.
* Parents or legal guardians provide informed consent for participation.

Exclusion Criteria:

* Presence of other syndromes or developmental disorders.
* History of recent surgical interventions or procedures involving the lower limbs.
* Significant neurological or orthopedic conditions that may affect gait.
* Any contraindications for participation in physical activities as determined by the child's healthcare provider.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Cadence | Immediately before the intervention and immediately after the intervention on the same day
  The number of steps taken per minute.

SECONDARY OUTCOMES:
Stride Length | Immediately before the intervention and immediately after the intervention on the same day
  The distance covered in a single step, measured in meters
Step Time: The duration of each step, measured in seconds | Immediately before the intervention and immediately after the intervention on the same day
  The duration of each step, measured in seconds
Velocity: | Immediately before the intervention and immediately after the intervention on the same day
  The speed of walking, measured in meters per second.
Joint Amplitudes | Immediately before the intervention and immediately after the intervention on the same day
  The angles at which the hip, knee, and ankle joints move during each phase of the gait cycle, assessed in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data Sensitivity: Given that the study focuses on a vulnerable population (children with Autism Spectrum Disorder), there are heightened concerns regarding the misuse or misinterpretation of the data.